CLINICAL TRIAL: NCT00049972
Title: An Open Label Study Assessing Paxil CR (Paroxetine CR) in Patients With Major Depressive Disorder Who Discontinued Treatment With Selective Serotonin Reuptake Inhibitors or a Selective Serotonin/Norepinephrine Reuptake Inhibitor Due to Intolerability
Brief Title: Major Depressive Disorder Study In Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: SB29060.833
Record Dates: First submitted 2002-11-18; First posted 2002-11-19 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder Open-label discontinued
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Drug: paroxetine CR

SUMMARY:
A study to obtain safety and tolerability data

ELIGIBILITY:
Inclusion Criteria:

* Patient must have primary diagnosis of Major Depressive Disorder (MDD).
* Discontinued a selective serotonin reuptake inhibitor (SSRI)or serotonin-norepinephrine reuptake inhibitor (SNRI) regimen due to intolerability.
* Minimum time frame between last dose of previous antidepressant and initiation of study drug is one week.
* Maximum time frame between last dose of prior antidepressant and initiation of study drug is 2 months.

Exclusion Criteria:

* Patient has previously been treated with the study drug.
* Is experiencing an adverse event attributed to previous SSRI/SNRI use that has not been resolved at least one week prior to Baseline Visit.
* Has a history of seizure disorder.
* Has met criteria for substance abuse or dependence within 6 months prior to Baseline Visit.
* Currently using an antidepressant.
* Currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646
Dates: Start 2002-09; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who prematurely terminated treatment due to treatment emergent adverse events

SECONDARY OUTCOMES:
Recurrence rates of adverse events causing intolerability of previous SSRI/SNRI, Adverse event incidence rates, Mean change from baseline in the Beck Depression Inventory-II total score, Proportion of responsers based on teh CGI Global Improvement Item

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Chair — GlaxoSmithKline
Locations (66):
- United States (66):
  - GSK Clinical Trial Call Center, Birmingham, Alabama
  - GSK Clinical Trial Call Center, Fairfield, Alabama
  - GSK Clinical Trial Call Center, Mobile, Alabama
  - GSK Clinical Trial Call Center, Phoenix, Arizona
  - GSK Clinical Trial Call Center, Little Rock, Arkansas
  - GSK Clinical Trial Call Center, Anaheim, California
  - GSK Clinical Trial Call Center, Anaheim Hills, California
  - GSK Clinical Trial Call Center, Bellflower, California
  - GSK Clinical Trial Call Center, Cerritos, California
  - GSK Clinical Trial Call Center, Clovis, California
  - GSK Clinical Trial Call Center, Encino, California
  - GSK Clinical Trial Call Center, Petaluma, California
  - GSK Clinical Trial Call Center, Riverside, California
  - GSK Clinical Trial Call Center, Sacramento, California
  - GSK Clinical Trial Call Center, San Francisco, California
  - GSK Clinical Trial Call Center, Temecula, California
  - GSK Clinical Trial Call Center, Vista, California
  - GSK Clinical Trial Call Center, Colorado Springs, Colorado
  - GSK Clinical Trial Call Center, Wilmington, Delaware
  - GSK Clinical Trial Call Center, Boynton Beach, Florida
  - GSK Clinical Trial Call Center, Delray Beach, Florida
  - GSK Clinical Trial Call Center, Fort Myers, Florida
  - GSK Clinical Trial Call Center, Melbourne, Florida
  - GSK Clinical Trial Call Center, Miami, Florida
  - GSK Clinical Trial Call Center, Ocala, Florida
  - GSK Clinical Trial Call Center, Atlanta, Georgia
  - GSK Clinical Trial Call Center, Idaho Falls, Idaho
  - GSK Clinical Trial Call Center, Gurnee, Illinois
  - GSK Clinical Trial Call Center, Greenwood, Indiana
  - GSK Clinical Trial Call Center, Lafayette, Louisiana
  - GSK Clinical Trial Call Center, Lake Charles, Louisiana
  - GSK Clinical Trial Call Center, New Orleans, Louisiana
  - GSK Clinical Trial Call Center, Prince Frederick, Maryland
  - GSK Clinical Trial Call Center, Springfield, Massachusetts
  - GSK Clinical Trial Call Center, Excelsior Springs, Missouri
  - GSK Clinical Trial Call Center, Kansas City, Missouri
  - GSK Clinical Trial Call Center, Saint Charles, Missouri
  - GSK Clinical Trial Call Center, St Louis, Missouri
  - GSK Clinical Trial Call Center, Las Vegas, Nevada
  - GSK Clinical Trial Call Center, Reno, Nevada
  - GSK Clinical Trial Call Center, Blackwood, New Jersey
  - GSK Clinical Trial Call Center, Mercerville, New Jersey
  - GSK Clinical Trial Call Center, Princeton, New Jersey
  - GSK Clinical Trial Call Center, Carrboro, North Carolina
  - GSK Clinical Trial Call Center, Cary, North Carolina
  - GSK Clinical Trial Call Center, Cincinnati, Ohio
  - GSK Clinical Trial Call Center, Cleveland, Ohio
  - GSK Clinical Trial Call Center, Independence, Ohio
  - GSK Clinical Trial Call Center, Oklahoma City, Oklahoma
  - GSK Clinical Trial Call Center, Eugene, Oregon
  - GSK Clinical Trial Call Center, Downingtown, Pennsylvania
  - GSK Clinical Trial Call Center, Bartlett, Tennessee
  - GSK Clinical Trial Call Center, Cordova, Tennessee
  - GSK Clinical Trial Call Center, Selmer, Tennessee
  - GSK Clinical Trial Call Center, Conroe, Texas
  - GSK Clinical Trial Call Center, Corsicana, Texas
  - GSK Clinical Trial Call Center, Dallas, Texas
  - GSK Clinical Trial Call Center, DeSoto, Texas
  - GSK Clinical Trial Call Center, Fort Worth, Texas
  - GSK Clinical Trial Call Center, Galveston, Texas
  - GSK Clinical Trial Call Center, Richardson, Texas
  - GSK Clinical Trial Call Center, Sugar Land, Texas
  - GSK Clinical Trial Call Center, West Valley City, Utah
  - GSK Clinical Trial Call Center, Lebanon, Virginia
  - GSK Clinical Trial Call Center, Richmond, Virginia
  - GSK Clinical Trial Call Center, Kirkland, Washington